CLINICAL TRIAL: NCT01395875
Title: Outcomes for Chronic Obstructive Pulmonary Disease Moderate Exacerbators Initiating Treatment
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113901
Record Dates: First submitted 2011-07-14; First posted 2011-07-18 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone-Salmeterol Drug Combination; Cholinergic Antagonists; Tiotropium Bromide; Ipratropium; Albuterol, Ipratropium Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COPD patients with moderate exacerbations: COPD patients with COPD-related using ICD-9 codes physician office/outpatient visit with a dispensing for oral corticosteroid (OCS) or antibiotic (ABX) within 5 days of the visit (Phy+Rx)
  Interventions: Drug: Fluticasone Propionate / Salmeterol Xinafoate Combination (FSC); Drug: Anticholinergics (AC)

INTERVENTIONS:
Drug: Fluticasone Propionate / Salmeterol Xinafoate Combination (FSC) — COPD patients receiving fluticasone propionate/salmeterol xinafoate combination (FSC) 250/50mcg
  Other Names: Advair (TM)
Drug: Anticholinergics (AC) — COPD patients receiving anticholinergics (ACs) including tiotropium (TIO) and ipratropium or combination ipratropium-albuterol (collectively referred to as ipratropium [IPR]).
  Other Names: Spiriva (TM); Atrovent (TM); Combivent (TM)

SUMMARY:
Patients with moderate COPD as defined by GOLD guidelines constitute almost 46% to 54% of all diagnosed COPD patients. Yet limited data exists on characterizing this study population in terms of drug therapy patterns and COPD-related resource use and costs. The objective of the following study was to conduct an analysis in the real-world setting to (1) identify and characterize COPD patients with moderate exacerbations and (2) evaluate the impact of initiating different maintenance therapies in this population. Maintenance therapy medications include inhaled corticosteroids (ICS), long-acting beta agonists (LABAs), combination of ICS+LABA, and anticholinergics (ACs) including tiotropium (TIO) and ipratropium or combination ipratropium-albuterol (collectively referred to as ipratropium [IPR]).

DETAILED DESCRIPTION:
Data from January 1, 2003 to March 31, 2009 will be available and termed as the study period. Patients with at least one moderate exacerbation defined as a physician/outpatient visit with a primary diagnosis of COPD and having an oral corticosteroid (OCS) or antibiotic prescription (ABX) within 5 days of physician/outpatient visit will be identified as the target population. The date of the first moderate exacerbation will serve as the patient's index date, and will be identified during the identification period of January 1, 2004 through February 28, 2009. Furthermore this moderate exacerbation should be the first medical claim with a primary diagnosis of COPD to ensure that only patients with moderate exacerbations will be captured. Subsequently, patients will be categorized into study cohorts based on the first maintenance drug prescription (index drug) received during the 30-day period after the index date termed as the treatment assessment period. Maintenance drugs considered include fluticasone-salmeterol 250/50 mcg (FSC) or anticholinergics (AC) including tiotropium (TIO) and ipratropium or combination ipratropium-albuterol (collectively referred to as ipratropium [IPR]). Patients not receiving any maintenance medication or those receiving maintenance medications other than those considered during the treatment assessment period will be excluded.

All outcomes will be assessed during a follow-up period that will vary in length between 1 day and 1 year for each patient. The variable follow-up period will be defined as the period that starts on the day after the treatment assessment period, and ends on the earliest of the following event dates: the end of the study period (March 31, 2009), the end of the patient's continuous eligibility in the health plan, the end of the patient's 1-year follow-up, treatment switch date (ie, a switch to any study medication different from the index drug), discontinuation date of the index drug (ie, more than a 60-day gap between the end of the days' supply of the preceding prescription and the fill date of the next consecutive prescription), or occurrence of any COPD-related exacerbation (COPD-related hospitalization, ED visit, or physician/outpatient visit with a prescription for an oral corticosteroid or antibiotic within 5 days of the visit).

A 1-year period before the index date (pre-period) will be used to provide a baseline assessment of the study cohorts. The specific dates for the pre- and follow-up periods will vary for each patient depending on their index date.

Specifically the study hypothesis for the primary outcome being tested was:

Ho: There is no difference in risk of any COPD-related exacerbation between FSC and AC cohorts Ha: There is a difference in risk of any COPD-related exacerbation between FSC and AC cohorts

Hypothesis for the key secondary outcome of COPD-related costs that was tested was:

Ho: There is no difference in COPD-related costs between FSC and AC cohorts Ha: There is a difference in COPD-related costs between FSC and AC cohorts

ELIGIBILITY:
Inclusion Criteria:

* minimum age 40 years at index
* continuously enrolled in health plan
* diagnosis of COPD (ICD-9 codes of 491, 492, 496)
* at least one moderate exacerbation event as defined previously.

Exclusion Criteria

* Exclusionary comorbid conditions of respiratory cancer, cystic fibrosis, fibrosis due to tuberculosis (TB), bronchiectasis, pneumonociosis, pulmonary fibrosis, pulmonary TB, or sarcoidosis
* Patients excluded if they did not receive treatment within the treatment assessment period following moderate exacerbation
* Receipt of maintenance medication in the pre-period
* Presence of treatment switch, discontinuation of index drug, or any COPD-related exacerbation during the treatment assessment period

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data from January 1, 2003 to March 31, 2009 will be available and termed as the study period. Patients with at least one moderate exacerbation defined as a physician/outpatient visit with a primary diagnosis of COPD (ICD-9 diagnosis codes) and having an oral corticosteroid (OCS) or antibiotic (ABX) prescription within 5 days of physician/outpatient visit will be identified as the target population. The date of this first moderate exacerbation will serve as the patient's index date, and will be identified during an identification period of January 1, 2004 to March 31, 2008 allowing for a maximum of a 1-year period before (pre-period) and after the index date (follow-up). The specific dates for the pre- and follow-up periods will be different for each patient depending on their index date. Furthermore this index moderate exacerbation should be the first medical claim with a primary diagnosis of COPD to ensure that only patients with moderate exacerbations will be captured.
Sampling Method: Non-Probability Sample
Enrollment: 2849 (Actual)
Dates: Start 2011-03; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
risk of any COPD-related exacerbation | January 1, 2003 to March 31, 2009 (up to 6 years)
  risk of the following types of COPD-related exacerbations between patients receiving FSC vs AC: COPD-related physician office/outpatient visit with a dispensing for oral corticosteroid (OCS) or antibiotic (ABX) within 5 days of the visit (Phy+Rx) and/or COPD-related hospitalization or an ED visit

SECONDARY OUTCOMES:
Moderate COPD exacerbation | January 1, 2003 to March 31, 2009 (up to 6 years)
  Risk of COPD-related exacerbations for patients with physician office/outpatient visit with a dispensing for oral corticosteroid (OCS) or antibiotic (ABX) within 5 days of the visit (Phy+Rx).
COPD-related hospitalization/ED | January 1, 2003 to March 31, 2009 (up to 6 years)
  Risk of COPD-related exacerbations for patients with COPD hospitalization with primary diagnosis code for COPD and ED visits with the same.
COPD-related Costs | January 1, 2003 to March 31, 2009 (up to 6 years)
  Comparing average monthly COPD-related costs and cost components between patients receiving FSC vs AC. Medical, pharmacy and total costs were examined

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline